CLINICAL TRIAL: NCT06201195
Title: Contribution of Anterior Femoral Cutaneous Nerve Block to Postoperative Analgesia for Total Knee Replacement
Brief Title: Anterior Cutaneus Nerve and Distal Adductor Canal Block With USG for Total Knee Replacement Analgesia
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Diskapi Teaching and Research Hospital (Other)
Responsible Party: Principal Investigator, derya özkan, professor, Diskapi Teaching and Research Hospital
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Supportive Care
Other Study IDs: AEŞH-EK1-2023-556
Record Dates: First submitted 2023-10-25; First posted 2024-01-11 (Actual); Last update posted 2025-11-19 (Actual); Status verified 2025-11

CONDITIONS: Pain Measurement; Knee Replacement Arthroplasty; Nerve Block
Keywords: anterior femoral cutaneus nerve block; distal adductor canal block; total knee arthroplasthy

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Adductor canal block (Active Comparator): Usg guidance adductor canal block with %0.25 Bupivacaine 20 ml
  Interventions: Procedure: Adductor canal blockade
- Distal adductor canal block with anterior cutaneus nerve block (Active Comparator): Usg guidance distal adductor canal block (%0.25 Bupivacaine 20 ml) with anterior cutaneus nerve block (%0.25 Bupivacaine 10 ml)
  Interventions: Procedure: Distal adductor canala blockade and anterior cutaneus nerve blockade

INTERVENTIONS:
Procedure: Adductor canal blockade — VAS, VAS move, incision place pain for up and down to patella, drain place pain, motor strenght for femoral nerve and siyatic nerve muscles, side effects, first analgesic requirement time, opioid requirement, other analgesics
  Other Names: first control
  Arms: Adductor canal block
Procedure: Distal adductor canala blockade and anterior cutaneus nerve blockade — VAS, VAS move, incision place pain for up and down to patella, drain place pain, motor strenght for femoral nerve and siyatic nerve muscles, side effects, first analgesic requirement time, opioid requirement, other analgesics
  Other Names: study group
  Arms: Distal adductor canal block with anterior cutaneus nerve block

SUMMARY:
This prospective clinical study was approved by the institutional ethics committee on September 27, 2023, and patient enrollment started in October 2023. the study aimed to evaluate the contribution of anterior femoral cutaneus nerve block to postoperative analgesia in total knee artroplasty.

The goal of this clinical trial is to compare analhesia effects of adductor canal blockade versus distal adductur canal blockade added anterior cutaneus nerve block in total knee arthroplasty.

The main questions it aims to answer are:

* question 1: does distal adductor canal blockade + anterior cutaneus nerve blokade superior analgesia then adductor canal block for undergoing TKP?
* question 2: does distal adductor canal blockade + anterior cutaneus nerve blokade decrease drain place pain on anterolateral face of knee?

DETAILED DESCRIPTION:
Patients with American Society of Anesthesiologists classification status I-III scheduled for elective primary TKA using standard spinal anesthesia enroll for this trial. After surgery patient divided two groups: 1- adductor canal blockade 2- distal adductor canal blockade + anterior femoral cutaneus nerve blockade. At postoperative 3th, 10th, 24th hour VAS (visuel analouge scale), VAS move, incision plase pain-for top and down of patella, drain place pain, motor strenght for femoral nerve and siyatic nerve, first analjesic requirement time, opioid consumption, total analcesic requirement will be recorded.

ELIGIBILITY:
Inclusion Criteria:

* Total knee artroplasty
* Spinal anesthesia
* ASA 1-3

Exclusion Criteria:

* Bupivacaine allergy
* Coagulopathy
* Infection on injection site

Ages: 40 Years to 85 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 58 (Actual)
Dates: Start 2023-10-01 (Actual); Primary Completion 2024-03-31 (Actual); Study Completion 2024-06-30 (Actual)

PRIMARY OUTCOMES:
VAS (visuel analouge scale) | postblock 3 hour,10 hour, 24 hour
  for postoperative pain evaluation after TKA surgery. The visual analogue scale (VAS) uses a 10 cm line with endpoint descriptors such as 'no pain' marked at the left end of the line and 'worst pain imaginable' marked at the right end.
drain place pain | postblock 3 hour,10 hour, 24 hour
  do you have any pain on drain place? yes or no

SECONDARY OUTCOMES:
VAS movement | postblock 3 hour,10 hour, 24 hour
  Postoperative pain with knee moves evaluate with VAS, The visual analogue scale (VAS) uses a 10 cm line with endpoint descriptors such as 'no pain' marked at the left end of the line and 'worst pain imaginable' marked at the right end.
motor strenght | postblock 3 hour,10 hour, 24 hour
  leg elevation and plantar flexion

CONTACTS AND LOCATIONS:
Overall Officials: Derya Ozkan, Study Director — Study Principal Investigator Ankara Etlik City Hospital; Müge Çakırca, doctor, Principal Investigator — Study Principal Investigator Ankara Etlik City Hospital; Funda Atar, doctor, Study Chair — Study Principal Investigator Ankara Etlik City Hospital; Serhan ünlü, doctor, Study Chair — Study Principal Investigator Ankara Etlik City Hospital
Locations (1):
- Ankara Etlik City Hospital, Ankara, Turkey (Türkiye)

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Bjorn S, Nielsen TD, Moriggl B, Hoermann R, Bendtsen TF. Anesthesia of the anterior femoral cutaneous nerves for total knee arthroplasty incision: randomized volunteer trial. Reg Anesth Pain Med. 2019 Dec 10:rapm-2019-100904. doi: 10.1136/rapm-2019-100904. Online ahead of print. PMID 31826920